CLINICAL TRIAL: NCT03676465
Title: CloudConnect: Predictive And Retrospective Clinical Decision Support For Chronic Disease Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Principal Investigator, Mark D. DeBoer, MD, MSc., MCR, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20958; 5R01LM012090 (NIH)
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Results first posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus (T1D); Continuous Glucose Monitor (CGM); Activity Monitor (i.e. Fitbit); Hemoglobin A1c (HbA1c); Companion Medical inPen; Insulin Pump; Multiple Daily Injections (MDI)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Subjects (child/parent dyad, with child and parent counted as separate subjects randomized together) will be randomized to either a Control Group or an Experimental Group. Both groups will use a study CGM and activity tracker. MDI users will use an inPen to dispense their insulin treatment with their personal insulin. Subjects who use an insulin pump to care for their diabetes will use their personal pump and their personal insulin during the study. All subjects will be asked to download their equipment each week. The study team will communicate with both the subject and their parent(s) each week to discuss their diabetes management. Subjects will complete questionnaires at the beginning and end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Subjects will wear their personal pump (if appropriate), use a study insulin pen (if appropriate), a study CGM and study activity tracker (i.e. Fitbit). Participants will receive a weekly CloudConnect Report based on analysis of the weekly data gathered for each participant. The report will be sent via email once a week to both the subject and their parent(s). Subjects and parents will have weekly contact with the study team. Subjects will complete questionnaires at the beginning and end of the study. These questionnaires will ask subjects about:
  * the communication within the family about the information shared in this report
  * how subjects feel when blood sugar is high or low
  * who takes responsibility of how diabetes care is managed
  Interventions: Other: CloudConnect Report
- Control Group (Active Comparator): Subjects will wear their personal pump (if appropriate), use a study insulin pen (if appropriate), a study CGM and study activity tracker (i.e. Fitbit). Participants will not receive a CloudConnect Report. Subjects and parents will have weekly contact with the study team. Subjects will complete questionnaires at the beginning and end of the study. These questionnaires will ask subjects about:
  * the communication within the family about the information shared in this report
  * how subjects feel when blood sugar is high or low
  * who takes responsibility of how diabetes care is managed
  Interventions: Other: Will not receive a CloudConnect Report

INTERVENTIONS:
Other: CloudConnect Report — Subjects and their parents will be asked to download the data from the study devices as well as download their insulin pump/pen. The participants will receive a weekly CloudConnect Report that is based on analysis of the data gathered from the downloads provided by the subject during that week. Participants will both receive weekly contact from the study team to discuss the communication that the subject & their parent had during the week about the participant's diabetes management.
  Arms: Experimental Group
Other: Will not receive a CloudConnect Report — Subjects and their parents will be asked to download the data from the study devices as well as download their insulin pump/pen. Participants will receive weekly contact from the study team to discuss the communication that the subject & their parent had during the week about the participant's diabetes management.
  Arms: Control Group

SUMMARY:
This study is to assess an approach of self-management called CloudConnect, evaluating the impact of CloudConnect Reports on patient engagement, adolescent/parent discussion, and clinical outcomes in adolescent Type 1 Diabetes (T1D).

DETAILED DESCRIPTION:
It is hypothesized that in contrast to adolescents randomized to the Control Group subjects will maintain a Hemoglobin A1c (HbA1c) while adolescents randomized to receiving the CloudConnect Report will have a lowering of HbA1c that is related to the increase in adolescent/parent disease-specific engagement. Moreover, the hypothesis is that the subjects receiving the CloudConnect Report will increase the engagement of adolescents/ parent through increased communication and self-management behavior, and that this increase in engagement will lead to improved medical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide informed consent
* Adolescents ages ≥12 and ≤ 17 years old with a parent/guardian (18+ yo) who is willing to participate with the child
* HbA1c ≥7 and ≤ 11 % (point-of-care machine or local laboratory [i.e. LabCorp]) (*This criteria only applies to the Main Study, it does not apply to the Pilot Study*)
* Willingness and ability to comply with scheduled visits and study procedures
* Willingness to comply with all the study devices during the entire trial (i.e. commercially-available CGM, Fitbit, Companion Medical inPen)
* One month stability on insulin parameters prior to enrollment
* MDI users should use Humalog® and Novolog® insulin to use in study insulin pen
* Type 1 diabetes mellitus diagnosed at least one year prior to enrollment in the study as noted by the following:

Criteria for documented hyperglycemia (at least 1 criterion must be met):

* Fasting glucose ≥ 126mg/dL-confirmed
* Two-hour Oral Glucose Tolerance Test (OGTT) ≥200mg/dL-confirmed hemoglobin A1c (HbA1c) ≥6.5% and documented by history - confirmed Random glucose ≥200 mg/dL with symptoms
* No data at diagnosis is available but the participant has a convincing history of hyperglycemia consistent with diabetes

Criteria for requiring insulin at diagnosis (at least 1 criterion must be met):

* Participant required insulin at diagnosis and continually thereafter
* Participant did not start insulin at diagnosis but upon investigator review likely needed insulin (significant hyperglycemia that did not respond to oral agents) and did require insulin eventually and used continually)
* The diagnosis of type 1 diabetes mellitus does not require documentation of C-peptide level or islet cell antibody positivity.
* Commitment to maintaining uninterrupted availability via cell phone at all times
* No diabetes complications
* Participants must demonstrate English proficiency and proper mental status and cognition for completion of the study.

  * Not currently known to be pregnant, breast feeding, or intending to become pregnant (females). A negative urine pregnancy test will be required for adolescent girls who are able to become pregnant. Participants who become pregnant will be discontinued from the study.
  * Ability to access the Internet to provide data to the clinical team or to travel to the research center so that the study equipment can be downloaded.
  * Medication stability in the preceding two months if taking antihypertensive, thyroid, anti-depressant or lipid lowering medication.

Exclusion Criteria:

* Children outside the ages of 12-17 y.o. or those who do not have a parent/guardian willing to participate
* Diabetic ketoacidosis in the past 6 months
* Pregnancy, breast-feeding, or intention of becoming pregnant
* Current or recent alcohol or drug abuse by patient history
* Mental incapacity, unwillingness or language barriers precluding adequate understanding, cooperation, or ability to fill out questionnaires.
* Any skin condition that prevents sensor placement (e.g., bad sunburn, pre-existing dermatitis, intertrigo, psoriasis, extensive scarring, cellulitis)
* Psychiatric disorders that would interfere with study tasks (e.g. cognitive disability, psychiatric hospitalization within 12 months)
* Use of acetaminophen (*this criteria only applies when the CGM version being used is older than the G6*)
* Use of long-acting insulin that is not Lantus or Tresiba
* For subjects who currently use a close-loop insulin pump and CGM: not being willing to turn off the closed-loop function
* Conditions that would make use of a CGM difficult (e.g., blindness, severe arthritis, immobility)
* Cystic fibrosis
* Current use of oral/inhaled glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study
* Any other comorbidity that at the judgment of the investigator may interfere with the participation on the study (i.e. uncontrolled high blood pressure or thyroid disease, current diabetic microvascular complications, current diagnose of gastroparesis)
* Severe hypoglycemia resulting in seizure or loss of consciousness in the 6 months prior to enrollment
* Use of a device that may pose electromagnetic compatibility issues and/or radiofrequency interference with the Dexcom CGM (implantable cardioverter-defibrillator, electronic pacemaker, neurostimulator, intrathecal pump, and cochlear implants)
* Active enrollment in another clinical trial

No eligiblity criteria is required for parent(s)/guardian(s) other than the legal relationship and 18+ yo.

List any restrictions on use of other drugs or treatments.

o Use of anti-diabetic agents other than short-acting insulin for CSII subjects or long-acting insulin for MDI subjects, including: metformin, sulfonylureas, meglitinides, thiazolidinediones, dipeptidyl peptidase 4 (DPP-4) inhibitors, glucagon-like peptide 1 agonists and alpha-glucosidase inhibitors

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D DeBoer, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeBoer MD, Valdez R, Corbett JP, Krauthause K, Wakeman CA, Luke AS, Oliveri MC, Chernavvsky DR, Patek SD. Effect of an Automated Advice Algorithm (CloudConnect) on Adolescent-Parent Diabetes-Specific Communication and Glycemic Management: A Randomized Trial. Diabetes Ther. 2023 May;14(5):899-913. doi: 10.1007/s13300-023-01401-9. Epub 2023 Apr 7. PMID 37027118

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From to 18 January 2019 to 13 January 2021, we a total of 132 participants (66 adolescent+parent dyads, each counted separately as participants) signed consent. Participants were recruited from the UVa Center for Diabetes Technology database and local Pediatric Endocrinology clinics.
Pre-assignment Details: 38 participants (19 adolescent+parent dyads) dropped out prior to randomization.
Units Other Than Participants: adolescent+parent dyad
Groups:
- Experimental Group: Subjects will wear their personal pump (if appropriate), use a study insulin pen (if appropriate), a study CGM and study activity tracker (i.e. Fitbit). Participants will receive a weekly CloudConnect Report based on analysis of the weekly data gathered for each participant. The report will be sent via email once a week to both the subject and their parent(s). Subjects and parents will have weekly contact with the study team. Subjects will complete questionnaires at the beginning and end of the study. These questionnaires will ask subjects about:
  * the communication within the family about the information shared in this report
  * how subjects feel when blood sugar is high or low
  * who takes responsibility of how diabetes care is managed
  CloudConnect Report: Subjects and their parents will be asked to download the data from the study devices as well as download their insulin pump/pen. The participants will receive a weekly CloudConnect Report that is based on analysis of the data gathered from the downloads provided by the subject during that week. Participants will both receive weekly contact from the study team to discuss the communication that the subject & their parent had during the week about the participant's diabetes management.
- Control Group: Subjects will wear their personal pump (if appropriate), use a study insulin pen (if appropriate), a study CGM and study activity tracker (i.e. Fitbit). Participants will not receive a CloudConnect Report. Subjects and parents will have weekly contact with the study team. Subjects will complete questionnaires at the beginning and end of the study. These questionnaires will ask subjects about:
  * the communication within the family about the information shared in this report
  * how subjects feel when blood sugar is high or low
  * who takes responsibility of how diabetes care is managed
  Will not receive a CloudConnect Report: Subjects and their parents will be asked to download the data from the study devices as well as download their insulin pump/pen. Participants will receive weekly contact from the study team to discuss the communication that the subject & their parent had during the week about the participant's diabetes management.
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 42; 21 adolescent+parent dyad | 52; 26 adolescent+parent dyad
Completed | 42; 21 adolescent+parent dyad | 44; 22 adolescent+parent dyad
Not Completed | 0; 0 adolescent+parent dyad | 8; 4 adolescent+parent dyad

BASELINE CHARACTERISTICS:
Population: These data represent the adolescent participants in the trial. Data were not collected regarding the parent who participated in survey questionnaires.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Categorical [Count of Participants; unit: Participants] — data refer to adolescent participants
  Participants
    <=18 years | 21 | 22 | 43
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.8 (1.5) | 14.8 (1.8) | 14.8 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants] — data refer to adolescent participants
  Participants
    Female | 9 | 11 | 20
    Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — data refer to adolescent participants
  Participants
    Hispanic or Latino | 0 | 2 | 2
    Not Hispanic or Latino | 21 | 20 | 41
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — data refer to adolescent participants
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 0 | 1
    White | 20 | 22 | 42
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: adolescents]
  United States | 21 | 22 | 43
Family Communication Inventory, Frequency scale [Mean (Standard Deviation); unit: units on a scale: FCI, Frequency] — The Family Communication Inventory, Frequency scale assesses the amount of times a parent and adolescent communicate regarding insulin dosing. Scores range from 0 to 36, with higher scores reflecting more frequent communication.
  units on a scale: FCI, Frequency | 12.0 (4.8) | 12.2 (7.3) | 12.1 (6.2)

OUTCOME MEASURES:

1. Primary Outcome: Family Communication Inventory Questionnaire
Description: It is hypothesized that individuals randomized to the Control Group will initially modestly improve management as a result of either of new access to CGM, but it will return to baseline levels by the 12-week evaluation. By contrast, it is hypothesize that individuals randomized to the Experimental Group will benefit from receiving the weekly CloudConnect Report by having increased engagement and communication by 8 weeks that is sustained by 12 weeks (3 months). The communication will be measured by comparing pre- and post-study Family Communication Inventory questionnaire and the weekly communication assessments. The Family Communication Inventory, Frequency scale assesses the amount of times a parent and adolescent communicate regarding insulin dosing. Scores range from 0 to 36, with higher scores reflecting more frequent communication--commonly thought of as a better outcome.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 21 | 22
Score on a scale | 12.3 (3.8) | 11.5 (6.7)
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Superiority; p > 0.05, t-test, 2 sided — Calculated p value was >0.05

2. Secondary Outcome: Glucose Time in Range 70-180 mg/dL, Overall
Description: Percentage of time during the study with glucose value between 70-180 mg/dL as measured by continuous glucose monitor, CGM
Time Frame: Overall (12 weeks)
Measure: Mean (Standard Deviation); unit: percentage of time in range 70-180 mg/dL
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 21 | 22
percentage of time in range 70-180 mg/dL | 47.6 (12.7) | 40.4 (7.5)
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Superiority; p > 0.05, t-test, 2 sided — Calculated p value was >0.05

3. Secondary Outcome: HbA1c, Final
Description: Final HbA1c measure
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: % of Hb
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 21 | 22
% of Hb | 7.58 (0.94) | 7.71 (1.11)
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Superiority; p > 0.05, t-test, 2 sided — Calculated p value was >0.05

4. Secondary Outcome: Mean Glucose by CGM
Description: Average glucose level measured by CGM
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 21 | 22
mg/dL | 198.2 (28.2) | 201.0 (27.6)
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Superiority; p > 0.05, t-test, 2 sided — Calculated p value was >0.05

5. Secondary Outcome: Percent Time <70 mg/dL
Description: Percentage of time participant spent with blood glucose below 70 mg/dL
Time Frame: 12-week
Measure: Median (Inter-Quartile Range); unit: % of time
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 21 | 22
% of time | 1.1 [0.6 to 2.9] | 1.2 [0.7 to 2.5]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Superiority; p > 0.05, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Percent Time >180 mg/dL
Description: Percentage of time participant spent with blood glucose greater than 180 mg/dL
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: % of time
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 21 | 22
% of time | 53.6 (12.8) | 54.0 (12.8)
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Superiority; p > 0.05, t-test, 2 sided — Calculated p value was >0.05

7. Secondary Outcome: Low Blood Glucose Episodes Per Week
Description: The number of episodes of hypoglycemia experienced each week
Time Frame: 12-week
Measure: Median (Inter-Quartile Range); unit: episodes per week
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 21 | 22
episodes per week | 2.75 [1.8 to 6.35] | 3.3 [1.2 to 5.3]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Superiority; p > 0.05, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Family Conflict Scale
Description: Score on the survey entitled Family Conflict Scale, which assesses the amount of Type 1 diabetes-related conflict between an adolescent and parent. Scores range from 19 to 57, with higher scores reflecting a greater amount of conflict--a worse outcome.
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 21 | 22
score on a scale | 25.4 (4.1) | 24.4 (5.1)
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Superiority; p > 0.05, t-test, 2 sided — Calculated p value was >0.05

9. Secondary Outcome: Division of Diabetes Responsibilities Score
Description: Adolescents completed the Division of Diabetes Responsibilities survey assessing their degree of responsibilities for given Type 1 diabetes management tasks, with scores ranging from 6 to 30 and with higher scores representing the adolescent assuming more responsibilities--commonly thought of as a better outcome.
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 21 | 22
Score | 21.3 (3.1) | 23.1 (4.5)
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Superiority; p > 0.05, t-test, 2 sided — Calculated p value was >0.05

10. Secondary Outcome: Child Self Management Score
Description: Scores on the Child Self Management are an assessment of the frequency over the past week of omitting T1D-related tasks for insulin dosing, with scores ranging from 0 to 30 and with higher scores representing more missed T1D-related tasks--commonly thought of as a worse outcome.
Time Frame: 12-week
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 21 | 22
Score on a scale | 4 [3 to 9.5] | 4 [2 to 6]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Superiority; p > 0.05, Wilcoxon (Mann-Whitney) — Calculated p value was >0.05

11. Secondary Outcome: My-Q
Description: Adolescent responses to My-Q relate to Type 1 diabetes-related quality of life, with scores ranging from 27-135 and with higher scores indicating a higher quality of life--a better outcome.
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 21 | 22
Score on a scale | 93.5 (11.9) | 95.8 (10.7)
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Superiority; p > 0.05, t-test, 2 sided — Calculated p value was >0.05

12. Secondary Outcome: Weekly Diabetes Communication
Description: Adolescent response to the question: "During the past week, did you talk with your parents about your diabetes management?"
Time Frame: 12-week
Population: Reduced numbers reflect missing data from individual participants.
Measure: Mean (Standard Deviation); unit: Percent of weeks with positive response
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 20 | 21
Percent of weeks with positive response | 88 (32) | 89 (31)
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Superiority; p > 0.05, Wilcoxon (Mann-Whitney) — Calculated p value was >0.05

13. Secondary Outcome: Tone of Response
Description: Adolescent rating Tone of response, i.e. whether Type 1 diabetes-specific communication has an overall positive or negative tone; scores ranged from 1 to 5, with 1 being a very negative tone and 5 being a very positive tone--a better outcome.
Time Frame: 12-week
Population: Reduced numbers reflect missing data from individual participants.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 20 | 21
Score | 3.58 (0.90) | 3.84 (0.87)
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Superiority; p > 0.05, Wilcoxon (Mann-Whitney) — Calculated p value was >0.05

14. Secondary Outcome: Change of Insulin Parameters
Description: Adolescent responding to the question, "During the past week, did you change your insulin parameters?"
Time Frame: 12-week
Population: Reduced numbers reflect missing data from individual participants.
Measure: Mean (Standard Deviation); unit: Percent of weeks with positive response
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 20 | 21
Percent of weeks with positive response | 0.36 (0.48) | 0.12 (0.33)
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 12-weeks
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group (N=21) | Control Group (N=22)
hypoglycemic seizure (Nervous system disorders) | 0 (0) | 1 (1) — Participant received insulin for dinner but did not eat much. She then went to a store with her sister who reports that the CGM was alarming and participant said her glucose was in the 60s. While waiting to buy a drink, she collapsed with a seizure.

LIMITATIONS AND CAVEATS:
We did not recruit our target number of participants because of changes in diabetes management during the study, with an increase in use of closed-loop systems, which were an exclusion criterion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT03676465/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT03676465/ICF_001.pdf